CLINICAL TRIAL: NCT04184323
Title: SIRT1-1 Antagonist Therapy Before Embryo Transfer to Improve Endometrial Receptivity and Life Pregnancy Rates
Brief Title: SIRT-1 Antagonism for Endometrial Receptivity
Acronym: SAFER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BL5280
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2020-11

CONDITIONS: Endometriosis; Uterine Diseases; Endometrial Diseases; Infertility Unexplained; Infertility; Female, Nonimplantation
Keywords: endometriosis; SIRT1; Progesterone resistance
MeSH Terms: conditions — Endometriosis; Uterine Diseases; Infertility; Progesterone Resistance | interventions — 6-chloro-2,3,4,9-tetrahydro-1H-carbazole-1-carboxamide

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled comparison of SirT1 inhibitor treatment for implantation failure associated with endometriosis
Who Masked: Participant, Care Provider, Investigator
Masking Description: Drug and placebo will be prepared in color coded capsules. Randomization will be performed using computer-generated lists assigned sequentially upon recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EX-527 (Active Comparator): The drug will be administered daily for 5 days beginning with the start of progesterone therapy and ended 24 hours before embryo transfer
  Interventions: Drug: EX-527 (Selisistat)
- Placebo (Placebo Comparator): The placebo will be administered daily for 5 days beginning with the start of progesterone therapy and ended 24 hours before embryo transfer
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EX-527 (Selisistat) — EX-527 is a specific inhibitor of the histone deacetylase Sirtuin-1 (SirT1). It is being given to reverse the effects of endometriosis, namely progesterone resistance, that is thought to interfere with the establishment of pregnancy in women with endometriosis
  Other Names: SEN0014196
  Arms: EX-527
Drug: Placebo — We will use the same vehicle for producing the active drug such as maltose without any hormones or active components
  Arms: Placebo

SUMMARY:
Progesterone resistance is mediated through epigenetic modification through SirT1 activation and is thought to contribute to infertility and progression of endometriosis. Endometriosis is a leading cause of unexplained IVF failure secondary to inflammatory changes that induce SirT1. The current study is designed to investigate a small molecule inhibitor of SirT1, in the clinical setting of In Vitro Fertilization and Embryo Transfer. The SAFER trial will compare EX-527 to placebo in a randomized, double-blind trial. Primary endpoints include Live Birth Rate (LBR) and secondary outcomes include pregnancy rate (PR), miscarriage rate (MR) and implantation failure rate.

DETAILED DESCRIPTION:
The SAFER Trial will enroll women with unexplained failure after embryo transfer with euploid embryos. Subjects must have existing euploid embryos for transfer and test positive for SirT1 testing on endometrial biopsy. To qualify, they must be 18 to 40 years of age, have a normal uterine cavity, no serious systemic diseases (diabetes, lupus, cancer, etc) and be willing to be randomized to treatment with a SirT1 inhibitor, EX-527 or placebo. The medication will be provided and administered for 5 days prior to embryo transfer, after progesterone therapy is begun. The drug will be stopped 24 hr before embryo transfer. Standard protocols will be used including administration of progesterone, checking hCG 8 days after transfer, ultrasound monitoring of pregnancy and pregnancy outcomes recording, with Live Birth Rate (LBR) being the primary outcome of interest. We expect to enroll 30 women, with 15 subjects per arm. The goal of this study is to demonstrate efficacy for a specific inhibitor of SirT1 as a primary treatment of defects in endometrial receptivity due to endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Must test positive for SIRT1 on mid-luteal endometrial biopsy
* Prior failed embryo transfer with euploid embryos
* Have at least one euploid embryo for transfer

Exclusion Criteria:

* systemic illness affecting kidneys or liver; chronic headache or severe migraine
* Endometritis, hydrosalpinges, and known adenomyosis
* Uterine septum, uterine fibroids, endometrial polyps

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy is a required end point
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 9 months to 2 years
  The number of successful pregnancies ending in live birth at the conclusion of the study divided by the number of embryo transfers in each group

SECONDARY OUTCOMES:
Pregnancy rate | 9 months to 2 years
  The number of subjects with a demonstrated pregnancy based on elevated and sustained hCG levels divided by the number of embryo transfers per group
Miscarriage rate | 9 months to 2 years
  The number of sustained pregnancies lost divided by the number of pregnancies in each group

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Lessey, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The demographic data, group assignment, and outcome data for each subject will be shared with other researchers including embryo grade, stage, pregnancy results (pregnant, not pregnant, miscarriage, ongoing pregnancy, Live birth)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of the study that includes live birth data

REFERENCES:
- [Background] Westerberg G, Chiesa JA, Andersen CA, Diamanti D, Magnoni L, Pollio G, Darpo B, Zhou M. Safety, pharmacokinetics, pharmacogenomics and QT concentration-effect modelling of the SirT1 inhibitor selisistat in healthy volunteers. Br J Clin Pharmacol. 2015 Mar;79(3):477-91. doi: 10.1111/bcp.12513. PMID 25223836
- [Background] Yoo JY, Kim TH, Fazleabas AT, Palomino WA, Ahn SH, Tayade C, Schammel DP, Young SL, Jeong JW, Lessey BA. KRAS Activation and over-expression of SIRT1/BCL6 Contributes to the Pathogenesis of Endometriosis and Progesterone Resistance. Sci Rep. 2017 Jul 28;7(1):6765. doi: 10.1038/s41598-017-04577-w. PMID 28754906
- [Background] Likes CE, Cooper LJ, Efird J, Forstein DA, Miller PB, Savaris R, Lessey BA. Medical or surgical treatment before embryo transfer improves outcomes in women with abnormal endometrial BCL6 expression. J Assist Reprod Genet. 2019 Mar;36(3):483-490. doi: 10.1007/s10815-018-1388-x. Epub 2019 Jan 4. PMID 30610661
- [Background] Almquist LD, Likes CE, Stone B, Brown KR, Savaris R, Forstein DA, Miller PB, Lessey BA. Endometrial BCL6 testing for the prediction of in vitro fertilization outcomes: a cohort study. Fertil Steril. 2017 Dec;108(6):1063-1069. doi: 10.1016/j.fertnstert.2017.09.017. Epub 2017 Nov 7. PMID 29126613